CLINICAL TRIAL: NCT03232398
Title: Apixaban Versus Warfarin in Patients With Left Ventricular (LV) Thrombus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, RONNY ALCALAI, Director, Cardiac Care Unit, Hadassah Medical Organization
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hadassah 0607-16
Record Dates: First submitted 2017-07-16; First posted 2017-07-28 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Acute Myocardial Infarction; Left Ventricular Thrombosis; Anticoagulants and Bleeding Disorders
MeSH Terms: conditions — Hemostatic Disorders | interventions — apixaban; Warfarin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The primary efficacy endpoint will be the presence of LV thrombus as assessed be echocardiography after 3 months of treatment. Echocardiography images will be reviewed for the presence of LV thrombus by two experts who will be blinded to the study drug.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apixaban (Active Comparator): Apixaban Oral Tablet [Eliquis]
  Interventions: Drug: Apixaban Oral Tablet [Eliquis]; Drug: Warfarin
- Warfarin (Active Comparator): Warfarin - Vitamin K antagonist
  Interventions: Drug: Apixaban Oral Tablet [Eliquis]; Drug: Warfarin

INTERVENTIONS:
Drug: Apixaban Oral Tablet [Eliquis] — Apixaban 5 mg BID for 3 months. Apixaban 2.5-mg BID doses will be used in a subset of patients with two or more of the following criteria: an age of at least 80 years, a body weight of no more than 60 kg, or a serum creatinine level of 1.5 mg per deciliter (133 μmol per liter) or more. Patients with advanced renal failure (CrCl between 15 ml/min and 29 mi/min) will also receive 2.5 mg BID.
  Other Names: Eliquis
Drug: Warfarin — Dose-adjusted warfarin to achieve a target international normalized ratio (INR) of 2.0 to 3.0 for 3 months
  Other Names: Coumadin

SUMMARY:
Patients with acute ST-segment elevation myocardial infarction (STEMI) have an elevated risk of stroke, most of which are cardio-embolic in origin as a result of left ventricular (LV) thrombus formation. Anterior-wall location of a MI, in particular, can lead to the complications of LV aneurysm and/or thrombus, which some estimate occurs in approximately up to one-third of individuals within the first 2 weeks following an anterior MI.

In the absence of anti coagulation, the risk of embolization in patients with a documented LV thrombus has been reported to be between 10 and 15 percent [3]. Although there are no randomized trials evaluating the efficacy of anticoagulation in patients with an LV thrombus after MI, observational studies provide substantial supporting evidence for the recommendation to anticoagulate patients with documented LV thrombus in order to reduce the risk of embolization. The observation that most events occur within the first three months from the MI forms the basis for the recommendation that anticoagulant therapy should be started early and continued for at least three to six months after myocardial infarction. Currently the practice guidelines recommend anticoagulation after MI only in certain settings such as the presence of LV thrombus or atrial fibrillation. To date there are no data on the use of novel oral anticoagulants (NOACS) for stroke prevention in the setting of LV thrombus after acute MI.

The proposed aim of this randomized open label non inferiority clinical trial is to assess whether apixaban is as effective as VKA for the treatment of LV thrombus after acute ST segment elevation MI.

Population: Patients with evidence of LV thrombus as assessed by trans-thoracic echocardiography (TTE) 3 to 7 days post admission for acute ST-elevation MI

Intervention: The patients will be randomly assigned to treatment with apixaban or s.c enoxaparin 1mg/Kg BID followed by dose-adjusted warfarin to achieve a target international normalized ratio (INR) of 2.0 to 3.0 for 3 months.

The study Outcomes are the presence of LV thrombus as assessed be echo, major bleeding, and stroke or systemic embolism and death from any cause.

DETAILED DESCRIPTION:
Background and Study Rationale:

Patients with acute ST-segment elevation myocardial infarction (STEMI) have an elevated risk of stroke, most of which are cardio-embolic in origin as a result of left ventricular (LV) thrombus formation. The risk for stroke after myocardial infarction (MI) is estimated to be 44-fold higher within the first 30 days, and remains 2 to 3 times higher than expected during the subsequent 3 years. Anterior-wall location of a MI, in particular, can lead to the complications of LV aneurysm and/or thrombus, which some estimate occurs in approximately up to one-third of individuals within the first 2 weeks following an anterior MI [2].

In the absence of anti coagulation, the risk of embolization in patients with a documented LV thrombus has been reported to be between 10 and 15 percent. Although there are no randomized trials evaluating the efficacy of anti coagulation in patients with an LV thrombus after MI, observational studies provide substantial supporting evidence for the recommendation to anti coagulate patients with documented LV thrombus in order to reduce the risk of embolization. The observation that most events occur within the first three months from the MI forms the basis for the recommendation that anticoagulant therapy should be started early and continued for at least three to six months after myocardial infarction.

Treatment of myocardial infarction has evolved dramatically in the past 20 years, and the vast majorities of patients undergo early coronary intervention and receive dual anti platelet therapy (DAPT). As a result, anterior MI alone does not warrant anti coagulation without evidence of LV thrombus since the combination of oral anti coagulation with DAPT carries an increased risk of bleeding. Practice guidelines recommend anti coagulation after MI only in certain settings such as the presence of LV thrombus or atrial fibrillation [5].

Recently oral thrombin inhibitors and factor Xa inhibitors (terms as novel oral anticoagulants - NOACS) have been introduced for stroke prevention in patients with non-valvular atrial fibrillation [6-8]. These agents were shown to be at least as effective as Vitamin K antagonists (VKA) such as warfarin in prevention of systemic embolism, while having an improved safety profile with less risk of bleeding.

To date there are no data on the use of NOACS for stroke prevention in the setting of LV thrombus after acute MI. Consequently, the effectiveness and safety of anti coagulation therapy with these novel agents in patients with LV thrombus warrants further investigation. The devastating impact of a stroke after an MI on morbidity and mortality, and the increasing number of patients at risk because of improved post-MI survival, making the goal of prevention of post MI stroke a major public health concern. The proposed study aims to address this important clinical topic.

Objective:

To assess whether apixaban is as effective as VKA for the treatment of LV thrombus after acute ST segment elevation MI.

Design Randomized open label non inferiority clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients with evidence of LV thrombus as assessed by trans-thoracic echocardiography
* Acute MI in last 3 months prior to enrollment

Exclusion Criteria:

* Patients with contraindications for chronic anti coagulation
* Patients with severe renal failure (CrCl< 15 ml/min)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Presence and dimensions of Left ventricular thrombus (LV) as assessed by 2D echocardiography | 3 months
  The primary efficacy endpoint will be the presence of LV thrombus as assessed be echocardiography after 3 months of treatment with oral anti coagulation. Dimensions of the LV thrombus (if still present) will be compared to the thrombus dimensions at baseline.

SECONDARY OUTCOMES:
Stroke or systemic embolism | 3 months
  Clinically significant stroke or systemic embolism requiring hospitalization
Major bleeding | 3 months
  Major bleeding, according to the criteria of the International Society on Thrombosis and Haemostasis (ISTH)
All cause mortality | 3 months
  Death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Ronny Alcalai, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Witt BJ, Brown RD Jr, Jacobsen SJ, Weston SA, Yawn BP, Roger VL. A community-based study of stroke incidence after myocardial infarction. Ann Intern Med. 2005 Dec 6;143(11):785-92. doi: 10.7326/0003-4819-143-11-200512060-00006. PMID 16330789
- [Background] Fuster V, Halperin JL. Left ventricular thrombi and cerebral embolism. N Engl J Med. 1989 Feb 9;320(6):392-4. doi: 10.1056/NEJM198902093200610. No abstract available. PMID 2913497
- [Background] Vaitkus PT, Barnathan ES. Embolic potential, prevention and management of mural thrombus complicating anterior myocardial infarction: a meta-analysis. J Am Coll Cardiol. 1993 Oct;22(4):1004-9. doi: 10.1016/0735-1097(93)90409-t. PMID 8409034
- [Background] Granger CB, Alexander JH, McMurray JJ, Lopes RD, Hylek EM, Hanna M, Al-Khalidi HR, Ansell J, Atar D, Avezum A, Bahit MC, Diaz R, Easton JD, Ezekowitz JA, Flaker G, Garcia D, Geraldes M, Gersh BJ, Golitsyn S, Goto S, Hermosillo AG, Hohnloser SH, Horowitz J, Mohan P, Jansky P, Lewis BS, Lopez-Sendon JL, Pais P, Parkhomenko A, Verheugt FW, Zhu J, Wallentin L; ARISTOTLE Committees and Investigators. Apixaban versus warfarin in patients with atrial fibrillation. N Engl J Med. 2011 Sep 15;365(11):981-92. doi: 10.1056/NEJMoa1107039. Epub 2011 Aug 27. PMID 21870978
- [Background] Schulman S, Kearon C; Subcommittee on Control of Anticoagulation of the Scientific and Standardization Committee of the International Society on Thrombosis and Haemostasis. Definition of major bleeding in clinical investigations of antihemostatic medicinal products in non-surgical patients. J Thromb Haemost. 2005 Apr;3(4):692-4. doi: 10.1111/j.1538-7836.2005.01204.x. PMID 15842354